CLINICAL TRIAL: NCT02469129
Title: Positron Emission Tomography (PET) Imaging of Poly(ADP-Ribose) Polymerase (PARP) Activity in Cancer
Brief Title: PET Imaging of PARP Activity in Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201410102
Record Dates: First submitted 2015-06-01; First posted 2015-06-11 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: positron emission tomography (PET) imaging; poly(ADP-ribose) polymerase 1 (PARP1); [18F]FluorThanatrace ([18F]FTT); PARP1 inhibitors; cancer treatments
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dosimetry Studies Arm (Experimental): Twelve participants with cancer and eight healthy volunteers will be recruited first to undergo whole-body PET/CT imaging to determine the whole body dosimetry of [18F]FluorThanatrace.
  Interventions: Drug: [18F]FluorThanatrace
- Kinetic Studies Arm (Experimental): An additional 30 participants with cancer will undergo a 1-hour dynamic scan upon injection of [18F]FluorThanatrace to determine the kinetics of the tracer in tumors to correlate with tissue-based markers of PARP activity and to obtain metabolite information to help determine the best quantification approach for the PET images. When possible these subjects will also undergo 18F-FDG imaging for comparison to tumor metabolism
  Interventions: Drug: [18F]FluorThanatrace

INTERVENTIONS:
Drug: [18F]FluorThanatrace — For the Dosimetry Studies, 10 mCi of [18F]FTT will be injected intravenously, and participants will be placed in the following groups to be imaged with PET at the specified time points: 0 minute group--image at 0 and 120 min. after tracer injection; 30 minute group--image at 30 and 150 min. after tracer injection; 60 minute group--image at 60 and 180 min. after tracer injection; and 90 minute group--image at 90 and 210 min. after tracer injection.
  For the Kinetic Studies, 10 mCi of [18F]FTT will be injected intravenously, and a 60-minute dynamic PET scan will be obtained starting at the time of injection.
  Other Names: [18F]FTT

SUMMARY:
The purpose of this research study is to determine the feasibility of using positron emission tomography (PET) imaging technology to image cancer with [18F]FluorThanatrace ([18F]FTT), a new radioactive tracer compound that has been developed that images poly(ADP-ribose) polymerase 1 (PARP-1) activity.

DETAILED DESCRIPTION:
Poly(ADP-ribose) polymerase 1 (PARP1) is a deoxyribonucleic acid (DNA) repair enzyme that enables normal cell survival as well as certain cancers. Pharmaceutical companies have invested heavily in PARP1 inhibitor development because these agents can effectively treat certain cancers as single agents, thus sparing those patients from chemotherapy toxicities. However, clinical trials testing PARP1 inhibitors have demonstrated mixed results due to the inability to measure the degree of PARP1 inhibition in tumors reliably. Accurately measuring tumoral PARP1 activity levels before and after PARP1 inhibitor treatment will: (1) enable identification of patients whose tumors exhibit PARP activity and are therefore good candidates for PARP inhibitor therapy, and (2) confirm that adequate doses of PARP1 inhibitors are being administered to patients, thus improving dose selection for further study in clinical trials. Thus, noninvasive approaches for measuring tumoral PARP1 activity would have commercialization potential in not only supporting development of PARP1 inhibitors but also after Food and Drug Administration (FDA) approval to assess clinical PARP1 inhibitor treatment responses.

Inflammation also contributes to a number of diseases involving the lungs and other organs. Increasing evidence suggests that PARP1 may also play a central role in modulating immune inflammatory responses. Thus, the data from this trial will also be used to develop this approach for studying lung inflammatory responses.

A new radiolabeled compound, [18F]FluorThanatrace ([18F]FTT), has been generated which can be used to measure PARP1 activity noninvasively and quantitatively using positron emission tomography (PET). Our data in cancer models show that the uptake of our compound is specific for PARP1 activity and correlates with biochemically determined PARP1 activity. Additional preliminary data also suggests that decreased [18F]FTT uptake predicts tumor response to PARP inhibition with olaparib, a PARP1 inhibitor currently being evaluated in clinical trials. Therefore, the investigators are conducting this Phase 0 trial to develop [18F]FTT for clinical use in cancer patients.

To date, no biomarkers have been developed beyond genetic testing for breast cancer 1 and 2 (BRCA1/2) mutations that can aid in patient selection for treatment with PARP inhibition. Moreover, no technologies are available to monitor the efficacy of PARP inhibition. Our technology provides both a biomarker for patient selection as well as a means of monitoring PARP activity during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or older.
* Healthy volunteers without history of cardiopulmonary conditions requiring any treatment or medical intervention and who are not current smokers (Dosimetry Studies Arm only).
* Patients with biopsy-proven diagnosis of head and neck squamous cell cancer (HNSCC) or any histopathologic type of lung cancer or any other type of cancer that can be treated with platinum-based chemotherapy as first-line therapy (which includes but is not limited to ovarian, gastric, and pancreatic cancers).
* At least one tumor site that is at least 1 cm in the shortest transaxial diameter by computed tomography (CT) (Kinetic Studies Arm only; disease-free participants can be enrolled in the Dosimetry Studies Arm).

Exclusion Criteria:

* History of claustrophobia or other preventing condition that has previously or would interfere with completion of protocol specified imaging sessions.
* Inability to comprehend or unwillingness to follow instructions for the study procedures as called for by the protocol.
* Presence of an implanted device that is incompatible with CT scanning.
* Non-measurable disease (< 1 cm) by CT (Kinetic Studies Arm only; disease-free participants can be enrolled in the Dosimetry Studies Arm).
* Unable to lie in the PET/CT scanner for the time required for scanning, up to 1 hour and 15 min at a time and possibly with arms raised above the head for lung imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Whole body effective dose and doses to critical organs (in rems) of a 10 millicurie (mCi) injection of [18F]FTT | This outcome measure is assessed from the [18F]FTT PET scan performed at the 1-day study visit.

SECONDARY OUTCOMES:
[18F]FTT maximum standard uptake value (SUV) in tumors | This is measured from the [18F]FTT PET scan performed at the 1-day study visit.
Distribution volume ratio (DVR) of [18F]FTT in tumors by Logan plot analysis | This is measured from the [18F]FTT PET scan performed at the 1-day study visit.
PARP enzyme activity | This is measured from the [18F]FTT PET scan performed at the 1-day study visit.
% positive poly(ADP)ribosylated (PAR) cells by immunohistochemistry | This is measured from the scheduled 1-day clinically-indicated biopsy or resection occurring closest to the 1-day PET scan visit for cancer patients in the Kinetic Arm.

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh L Dehdashti, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States